CLINICAL TRIAL: NCT06999057
Title: Quadriceps Motor Unit Adaptation to Simulated Knee Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Grant Norte, Associate Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Knee_Injection_Study:6295
Record Dates: First submitted 2025-05-20; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Muscle Inhibition; Knee Injury Simulation
Keywords: Quadriceps; Electromyography; Motor Unit; Knee Effusion; Lidocaine; Deafferentation; Neuromuscular Adaptation; Muscle Strength
MeSH Terms: interventions — Lidocaine; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Effusion Group (Experimental): 60 mL sterile saline injected into knee
  Interventions: Device: Joint Effusion via 60 mL Sterile Saline
- Deafferentation Group (Active Comparator): Lidocaine (single intra-articular dose)
  Interventions: Drug: Intra-articular Lidocaine
- Control Group (Sham Comparator): Sham procedure with fake needle
  Interventions: Other: Sham injection

INTERVENTIONS:
Device: Joint Effusion via 60 mL Sterile Saline — Injection of sterile saline into the knee joint to simulate joint swelling and induce quadriceps inhibition.
  Arms: Effusion Group
Drug: Intra-articular Lidocaine — Injection of 7 mL lidocaine into the knee joint to simulate deafferentation by temporarily blocking sensory input.
  Arms: Deafferentation Group
Other: Sham injection — Simulated knee injection using a stage needle without skin penetration, used to blind participants and serve as control.
  Arms: Control Group

SUMMARY:
This study investigates how simulated knee injury-via artificial joint effusion or deafferentation-affects quadriceps motor unit behavior in healthy young adults. Participants will complete neuromuscular testing during a single 2-hour lab session. This research seeks to improve understanding of muscle inhibition and inform interventions after real-world knee trauma.

DETAILED DESCRIPTION:
Using a controlled laboratory model, the investigators will simulate knee injury through two methods: (1) intra-articular saline injection to induce effusion, and (2) intra-articular lidocaine injection to induce sensory deafferentation. Healthy participants aged 18-30 will undergo surface and decomposition EMG, isometric strength testing, and reflex measurements before and after the intervention. The primary outcome is motor unit recruitment characteristics, with secondary outcomes including quadriceps inhibition (Hoffmann reflex) and isometric peak torque. The findings will inform future neuromodulatory approaches in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-30 years
2. Physically active (Tegner ≥ 5)
3. No prior lower-limb surgery or major injury

Exclusion Criteria:

1. Lower limb surgery or significant injury in past 2 years
2. Cardiopulmonary, neurological, or psychiatric disorders
3. Needle/electrical stimulation anxiety
4. Medications affecting neuromuscular or psychological function
5. Pregnancy
6. Allergic to lidocaine
7. Inability to elicit Hoffmann reflex

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Motor Unit Recruitment (amplitude relative to recruitment threshold) | Baseline, 0, 30, and 60 minutes post-intervention
  Measured via surface EMG decomposition
Motor Unit Recruitment (firing rate relative to recruitment threshold) | Baseline, 0, 30, and 60 minutes post-intervention
  Measured via surface EMG decomposition

SECONDARY OUTCOMES:
Quadriceps Inhibition (Hoffmann Reflex) | Baseline, 0 and 60 minutes post-intervention
  Measured with femoral nerve stimulation
Isometric Peak Torque (Quadriceps Strength) | Baseline and 60 minutes post-intervention
  Measured with isokinetic dynamometer (Biodex)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes, including motor unit recruitment characteristics, quadriceps strength, and Hoffmann reflex measurements, will be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting documentation will be available beginning 6 months after publication of the primary manuscript. Data will remain available for 5 years following that date.
Access Criteria: Qualified researchers with appropriate data use agreements in place may request access. Requests should be submitted to the Principal Investigator via email and will be reviewed by the study team. Data will be shared via secure file transfer protocols.